CLINICAL TRIAL: NCT01363115
Title: Calcium Supplementation for a Healthy Weight (CaSHeW)
Acronym: CaSHeW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Beverage Institute for Health & Wellness (Other)
Responsible Party: Lee M. Kaplan, MD, PhD, Massachusetts Genral Hosptial
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-P-000414
Record Dates: First submitted 2011-05-26; First posted 2011-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Obesity; Overweight
Keywords: Body Weight; Dietary Supplement; Calcium; Vitamin D
MeSH Terms: conditions — Obesity; Overweight; Body Weight | interventions — Calcium; Vitamin D; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OJ fortified with Ca and VitD (Experimental): Regular OJ fortified with Calcium (350 mg/8 fluid oz serving) and Vitamin D3 (100 IU/8 fluid oz serving): one 8 fluid oz serving three times/day (treatment) in combination with nutritional counseling
  Interventions: Dietary Supplement: Orange Juice fortified with Calcium and Vitamin D; Behavioral: Nutritional Counseling
- OJ without VitD and Ca (Active Comparator): Regular OJ without Calcium or Vitamin D3: one 8 fluid oz serving three times/day (control)
  Interventions: Dietary Supplement: Orange juice without Ca or VitD; Behavioral: Nutritional Counseling

INTERVENTIONS:
Dietary Supplement: Orange Juice fortified with Calcium and Vitamin D — Three 240 mL glasses of orange juice fortified with 350 mg Ca and 100 IU of D per serving
  Other Names: Minute Maid regular calorie orange juice
  Arms: OJ fortified with Ca and VitD
Dietary Supplement: Orange juice without Ca or VitD — Three 240 mL glasses of orange juice without Ca or VitD
  Other Names: Minute Maid regular calorie orange juice
  Arms: OJ without VitD and Ca
Behavioral: Nutritional Counseling — Individual and group nutritional counseling by a registered dietitian

SUMMARY:
The objective of this study is to investigate the effect of calcium (Ca) and vitamin D (D) supplemented orange juice (OJ) on weight loss and visceral fat mass in overweight and obese adults.

DETAILED DESCRIPTION:
The prevalence of obesity and levels of overweight is rising worldwide. In the United States, 63% of men and 55% of women are now overweight or obese. Recent epidemiological data and clinical trials have shown that a small daily increase in calcium or dairy products may result in annual losses in body weight and body fat. Data from clinical studies suggest that a 1000 mg per day increase in calcium intake is associated with an 8 kg difference in mean body weight and that calcium intake explains about 3% of the variance in body weight.

The objective of this study is to investigate the effect of calcium (Ca) and vitamin D (D) supplemented orange juice (OJ) on weight loss and visceral fat mass in overweight and obese adults.

Otherwise healthy overweight and obese men and women ages 18 to 65 years with a BMI between 25 and 35 kg/m2 will be randomized into one of the following experimental groups (36 in each group):

1. Regular OJ: one 8 fluid oz serving three times/day (control)
2. Regular OJ fortified with Calcium (350 mg/8 fluid oz serving) and Vitamin D3 (100 IU/8 fluid oz serving): one 8 fluid oz serving three times/day (treatment)

Subjects will receive either orange juice (OJ) (control) or OJ fortified with calcium and vitamin D3 (treatment) for 16 weeks. The study will involve 6 outpatient study visits to the study center.

Primary endpoint: Change in body weight after 16 weeks Secondary endpoint: Visceral fat change after 16 weeks as measured by single slice CT scan

ELIGIBILITY:
Inclusion Criteria:

* Men or women, between 18 and 65 years of age, who are capable of providing informed consent.
* BMI of 25 to 35 kg/m2
* Non-smoker (for at least 6 months).
* In good health, as determined by the principal investigator based on medical history and physical examination.
* Clinical laboratory evaluations (including Biochemistry, Hematology, Urinalysis) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator.
* Because of the calorie-restricted diet and radiation exposure from the CT scan, females will be non-pregnant, non-lactating, and either post-menopausal for at least 1 year, surgically sterile for at least 3 months, or be willing to use an approved method of contraception (which may include use of abstinence; non-hormonal intrauterine device with spermicide; female condom with spermicide; diaphragm with spermicide; cervical cap with spermicide; oral or transdermal hormonal contraceptives; a condom with spermicide by the sexual partner; or a sterile sexual partner) from 35 days prior to study entry (i.e., Day -1) until 30 days following Study Completion. For all females, the pregnancy test result must be negative at the screening visit and at visits when a CT scan will be done.
* Ability to comprehend and willingness to sign the Informed Consent Form for this study.
* Ability to comply with study restrictions regarding diet and exercise
* Stable weight (+ 5%) for at least 3 months prior to study entry.

Exclusion Criteria:

* Diabetes mellitus
* History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders which in the opinion of the investigator would be expected to interfere with the study or increase risk to the subject.
* Participation in any other investigational diet study within 90 days prior to study entry.
* History of a medical or psychological condition or social circumstances that would impair the subject's ability to participate reliably in the study.
* Use within the last six months of medications that can result in significant weight gain or weight loss, including antipsychotics, selective serotonin reuptake inhibitors, anti-epileptic drugs, appetite-suppressants such as phentermine and sibutramine, and the lipase-inhibitor orlistat.
* Active eating disorder
* History of alcoholism or substance abuse within 5 years prior to study entry.
* Use of a dietary supplement or medication that decreases calcium absorption
* History of kidney stone, hyperparathyroidism or sarcoidosis
* High calcium intake (more than 2 servings of dairy products per day or taking calcium supplements > 3x/wk ) for 1 month prior to study start date and for duration of study. (If participant is taking calcium supplement > 3x/wk or more than 2 servings of dairy products per day, they are eligible to participate if they agree to stop for 1 month prior to study start date and for the duration of the study. Participants will similarly be asked to stop multivitamins as the majority of these supplements contain calcium.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-07; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline and 16 weeks

SECONDARY OUTCOMES:
Change in visceral adipose tissue mass | Baseline and 16 weeks
Change in subcutaneous adipose tissue mass | Baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Kaplan, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Weight Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Rosenblum JL, Castro VM, Moore CE, Kaplan LM. Calcium and vitamin D supplementation is associated with decreased abdominal visceral adipose tissue in overweight and obese adults. Am J Clin Nutr. 2012 Jan;95(1):101-8. doi: 10.3945/ajcn.111.019489. Epub 2011 Dec 14. PMID 22170363